CLINICAL TRIAL: NCT06159504
Title: Simplifying Hepatitis C Pathways for People Who Inject Drugs in Armenia, Georgia, and Tanzania (CUTTS HepC): a Non-randomised, Quasiexperimental, Prospective Comparative Trial
Brief Title: Simplifying Hepatitis C Pathways for People Who Inject Drugs in Armenia, Georgia, and Tanzania
Acronym: CUTTS HepC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Médecins du Monde (Other)
Collaborators: UNITAID (Other); Burnet Institute (Other); University of Bristol (Other); International Network of People who Use Drugs (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUTTS HepC / HCV MoC
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis C; RDT
Keywords: Point of care (PoC); Nucleic acid testing; Qualitative interviews; Feasibility; Acceptability; Cost-effectiveness; Modelling
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; velpatasvir

STUDY DESIGN:
Intervention Model Description: Two study groups will be running in tandem/parallel to one another at the same time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 - simplified care model (Active Comparator): Arm 1 will receive DAA medication at the second appointment following the return of RNA HCV results. They will receive sofosbuvir (400mg) and velpatasvir (100mg).
  Interventions: Drug: sofosbuvir/velpatasvir (SOF/VEL)
- Arm 2 - short read time (Experimental): Arm 2 will begin DAA treatment after the first appointment following a shortened RDT read time of 5 minutes rather than 20 minutes. They will receive sofosbuvir (400mg) and velpatasvir (100mg).
  Interventions: Drug: sofosbuvir/velpatasvir (SOF/VEL); Diagnostic Test: Shortened read time of rapid diagnostic test for hepatitis C virus.

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir (SOF/VEL) — 400mg of SOF and 100mg of VEL self administered daily as a tablet.
Diagnostic Test: Shortened read time of rapid diagnostic test for hepatitis C virus. — Administered once during hepatitis C testing. Test is read after 5 minutes rather than its usual time of 20 minutes.
  Other Names: OraQuick® HCV RDT
  Arms: Arm 2 - short read time

SUMMARY:
The goal of this non-randomised, quasi-experimental, prospective comparative trial is to trial simplified care pathways for hepatitis C testing and treatment for people who inject drugs in Armenia, Georgia, and Tanzania.

The main questions it aims to answer are:

1. What is the feasibility of implementing a hepatitis C simplified care and same-day treatment care model in community and harm reduction settings in the three study countries?
2. Does a same-day treatment initiation model involving only POC antibody tests (with a shortened read-time) increase hepatitis C treatment uptake and SVR12 outcome (cure) among people who inject drugs compared with a simplified care model involving POC antibody followed by a confirmatory RNA test?
3. What is the comparative cost-effectiveness between a same-day antibody only hepatitis C testing and treatment model and the simplified care model (POC antibody/confirmatory RNA test) model?

Participants will:

* be enrolled in a new simplified model of care in each country (Arm 1). After the enrolment target is met for Arm 1 (approx. 3-9 months into implementation) new participants will be enrolled into a same-day treatment trial, using presumptive treatment after a reactive POC test result at shortened read-time (5minutes) (Arm 2)
* if in Arm 1, participants will commence SOF-VEL DAA treatment after receiving an RNA test to confirm current hepatitis C infection. They will then continue along the treatment pathway, returning for RNA testing 4-16 weeks after SVR12 to determine cure.
* if in Arm 2, participants will begin SOF-VEL DAA treatment on the same day as the 5 minute RDT testing. They will then continue along the treatment pathway, returning for RNA testing 4-16 weeks after SVR12 to determine cure.

Researchers will compare cure and participant retention rates between the two groups.

DETAILED DESCRIPTION:
The investigators will conduct a study to trial a new, simplified, and lower cost clinical pathway and determine its feasibility, effectiveness, cost-effectiveness and acceptability in Armenia, Georgia, and Tanzania.

This is a non-randomised, quasi-experimental, prospective comparative trial with approximately 350 participants initiated onto hepatitis C treatment in each arm. Arm one is a simplified care model (following global guidance) with hepatitis C treatment commencing after a rapid hepatitis C antibody test and a confirmatory positive hepatitis C ribonucleic acid (RNA) test. Arm two will involve same day treatment commencement following a positive rapid antibody test without confirmatory RNA testing prior to treatment initiation (RNA testing will be completed after treatment is provided). In arm two, the decision to treat will be based on the result of an early read time (< 5 mins) of a rapid antibody test which previous research findings suggest correlates strongly with a hepatitis C RNA positive test result. All positive participants will be treated with sofosbuvir (400mg) and velpatasvir (100mg), self-administered orally once per day for 12 weeks. Hepatitis C cure will be assessed by sustained virological response (SVR) laboratory testing.

The first primary outcome is feasibility, measured throughout the care cascade. Primary outcomes compared across the two arms will be the proportion of participants 1) commencing treatment and 2) achieving SVR. Test concordance and validity of the early read time will be assessed against laboratory RNA test results (which will also guide decisions to continue or cease treatment in Arm 2). A mixed effects model will be used to assess study outcomes and infectious diseases modelling will determine cost-effectiveness. The acceptability and feasibility of the models will be assessed through thematic analysis of participant and practitioner interviews, and site assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able and willing to provide informed consent in local language
* Not currently on or previously had treatment for hepatitis C
* Attending site for needle / syringe program, OR self-reports ever injecting drugs

Exclusion Criteria:

* Self-reported history of decompensate cirrhosis of the liver
* Women who are pregnant or breast-feeding
* Self-report other significant co-morbidities such as uncontrolled HIV infection, history of renal dysfunction, tuberculosis infection, or chronic hepatitis B infection
* Unable / unwilling to stop any contraindicated medications / supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3040 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The feasibility of implementing a hepatitis C simplified care (Arm 1) and same-day treatment (Arm 2) care models in community and harm reduction settings in the three study countries. | 3 years
  Measured through case report forms, interviews and study site checks.
The proportion of participants initiating hepatitis C treatment in simplified care Arm vs same-day treatment Arm. | 3 years
The proportion of participants who achieve SVR following hepatitis C treatment in simplified care Arm vs same-day treatment Arm. | 3 years
The comparative cost and cost-effectiveness of simplified care vs same-day treatment models of care. | 3 years

SECONDARY OUTCOMES:
Participant acceptability of the hepatitis C simplified care and same-day treatment care models. | 3 years
  Measured through interviews and surveys
Practitioner acceptability of hepatitis C simplified care and same-day treatment care models | 3 years
  Measured through interviews
The time to treatment initiation among participants in simplified care Arm vs same-day treatment Arm | 3 years
The proportion of participants who complete hepatitis C treatment in simplified care Arm vs same-day treatment Arm | 3 years
The proportion of participants whose hepatitis C antibody test result at 5-min read-time concords with RNA test results. | 3 years
Identification of the optimal "cut-off" read-time for hepatitis C antibody test to predict RNA positivity | 3 years
The proportion of participants "overtreated" for hepatitis C in the same-day treatment Arm. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hellard, Principal Investigator — Burnet
Locations (1):
- National Institute for Infectious Diseases, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided